CLINICAL TRIAL: NCT04978636
Title: The eFfect of cOntinuous Low Tidal Volume Ventilation With Hyperoxia Avoidance During CardiopUlmonary Bypass "FOCUS" Trial Blood Samples
Brief Title: Low Tidal Volume Ventilation With Hyperoxia Avoidance During Cardiopulmonary Bypass (The FOCUS Trial)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Society of Cardiovascular Anesthesiologists (Unknown); University of Pittsburgh Medical Center (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Marta Kelava, MD, PI, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 21-447
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous low-tidal volume ventilation with using FiO2 of 0.21 (Active Comparator): The investigator will investigate the effect of continuous low tidal volume ventilation with hyperoxia avoidance (using FiO2 of 0.21) on PPCs and 30-day mortality compared to low-tidal volume ventilation (with FiO2 of 0.21) or apnea during CPB, and during the sub-study.
  Interventions: Other: Continuous low-tidal volume ventilation with using FiO2 of 0.21
- Continuous low tidal volume ventilation with using FiO2 of 1.0 (Active Comparator): The investigator will investigate the effect of low tidal volume lung ventilation with hyperoxia avoidance (FiO2 of 0.21) on PPCs and mortality compared to hyperoxic low-tidal volume ventilation (with FiO2 of 1.0) or apnea during CPB, and during the sub-study.
  Interventions: Other: Continuous low tidal volume ventilation with using FiO2 of 1.0
- Apnea (Active Comparator): The investigator will investigate the effect of apnea during on PPCs and mortality compared to hyperoxic low-tidal volume ventilation (with FiO2 of 1.0) or hyperoxia avoidance (FiO2 of 0.21) during CPB, and during the sub-study..
  Interventions: Other: Apnea During CPB

INTERVENTIONS:
Other: Continuous low-tidal volume ventilation with using FiO2 of 0.21 — The continuous low-tidal volume ventilation with using FiO2 of 0.21 will be defined as the tidal volume of 3 mL/kg IBW (up to maximum 200 mL), 0.21 of FiO2, respiratory rate of 5 per minute, and PEEP 5 cm H20). A recruitment maneuver with 30 cm H2O for 10 seconds will be performed before starting the selected ventilation mode in all patients. During the sub-study extra blood samples will be drawn before and after CPB.
  Arms: Continuous low-tidal volume ventilation with using FiO2 of 0.21
Other: Continuous low tidal volume ventilation with using FiO2 of 1.0 — The continuous low-tidal volume ventilation with using FiO2 of 1.0 will be defined as the tidal volume of 3 mL/kg IBW (up to maximum 200 mL), 1.0 of FiO2, respiratory rate of 5 per minute, and PEEP 5 cm H20). A recruitment maneuver with 30 cm H2O for 10 seconds will be performed before starting the selected ventilation mode in all patients. During the sub-study extra blood samples will be drawn before and after CPB.
  Arms: Continuous low tidal volume ventilation with using FiO2 of 1.0
Other: Apnea During CPB — There will be no ventilation used. But, during the sub-study part of the Apnea CPB extra blood samples will be drawn before and after CPB.
  Arms: Apnea

SUMMARY:
This is a multi-institutional study (CCF, UPMC, OSU) evaluating different ventilation strategies during cardiopulmonary bypass on mortality and postoperative pulmonary complications, with sub-study investigating 8-iso-prostaglandin F2a and sRAGE levels.

DETAILED DESCRIPTION:
The investigators will evaluate the effect of low tidal volume with varying FiO2 fractions during cardiopulmonary bypass on postoperative mortality and pulmonary complications. This will be a prospective, pragmatic, cluster randomized trial including all eligible adult cardiac surgical patients requiring cardiopulmonary bypass. Each week, all operating rooms will be randomized to one of three possible ventilation strategies during the period of cardiopulmonary bypass: 1) continuous low tidal volume ventilation with inspired oxygen fraction at 1.0, 2) continuous low tidal volume ventilation with inspired oxygen fraction at 0.21, and 3) no ventilation (apnea). The investigators will anticipate increase in plasma sRAGE and 8-iso-prostaglandin F2a levels in all three groups of patients during CPB with the highest levels immediately after cross-clamp release. The investigators will anticipate significant difference with at least 25% lower sRAGE levels in this group. The sub-study will also provide preliminary data on the behavior of the 8-iso-prostaglandin F2a which will be useful in further investigation of other targeted interventions to reduce ischemia-reperfusion injury to the lung during routine cardiac surgical operations.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Male and female patients undergoing elective cardiac surgeries requiring cardiopulmonary bypass.

Exclusion Criteria:

Emergency surgeries, surgeries requiring lung isolation and one-lung ventilation (OLV), heart or lung transplants, and mechanical circulatory support device implantation pulmonary thrombendarterectomies.

* Surgeries requiring one-lung ventilation will be excluded because of the inability to employ study intervention and the differential treatment of the lungs likely confounding any potential effect from the planned intervention.
* Lung transplant surgeries will be excluded for similar reasons as well as other confounding effects affecting the primary composite outcome.
* Heart transplants and mechanical circulatory support device implantation surgeries will be excluded because these patients already receive intervention as part of the institutional protocol at the primary study site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5502 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Composite including STS 30 day Mortality and postoperative pulmonary complications | Within 30 days of surgery
  Composite including STS 30-day mortality and postoperative pulmonary complications defined a early respiratory failure defined as PaO2/FiO2 ratio<200 mmHg at any time within the first 24 hours of ICU admission, postoperative reintubation during the hospital stay, prolonged ventilation, pneumonia, pleural effusion requiring drainage, pneumothorax requiring intervention, and readmission due to: pleural effusion requiring intervention, or pneumonia.

SECONDARY OUTCOMES:
CPB time | During surgery
  Duration of cardiopulmonary bypass (STS defined)
ICU LOS | Within 30 days of surgery
  ICU length of stay (STS defined)
Early respiratory failure - PaO2/FiO2 ratio < 200 mmHg at any time within the first 24 hours of ICU admission | 24 hours
  PaO2/FiO2 ratio < 200 mmHg at any time within the first 24 hours of ICU admission
Hospital LOS | Within 30 days of surgery
  Hospital length of stay (STS defined)
Reintubation | Within 30 days of surgery
  Reintubation (STS defined)
Need for tracheostomy | Within 30 days of surgery
  Need for tracheostomy (STS defined)
Pleural effusion requiring drainage | Within 30 days of surgery
  Pleural effusion requiring drainage (STS defined)
Pneumonia | Within 30 days of surgery
  Pneumonia (STS defined)
Readmission | within 30 days of surgery
  Readmission due to respiratory complication or need for thoracentesis and chest tube insertion (STS defined)
30-day mortality | Within 30 days of surgery
  STS defined in hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Marta Kelava, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States